CLINICAL TRIAL: NCT04250246
Title: A Randomized, run-in, Multi-center, Phase II Study of Nivolumab Combined With Ipilimumab and Guadecitabine or Nivolumab Combined With Ipilimumab in Melanoma and NSCLC Patients Resistant to Anti-PD-1/PD-L1 (NIBIT-ML1)
Brief Title: A Study of NIVO Plus IPI and Guadecitabine or NIVO Plus IPI in Melanoma and NSCLC Resistant to Anti-PD1/PDL1
Acronym: NIBIT-ML1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Italian Network for Tumor Biotherapy Foundation (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBIT-ML1
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Melanoma; Non Small Cell Lung Cancer
Keywords: melanoma; NSCLC; ipilimumab; nivolumab; guadecitabine
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Nivolumab; guadecitabine

STUDY DESIGN:
Intervention Model Description: Randomized, non-comparative, phase II study designed according to a two stages optimal design by Simon
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ipilimuamb plus nivoluamb plus guadecitabine (Experimental): ipilimumab plus nivolumab combined with guadecitabine
  Interventions: Drug: Ipilimumab plus nivolumab plus guadecitabine
- Ipilimumab plus nivolumab (Active Comparator): Ipilimumab plus nivolumab
  Interventions: Drug: Ipilimumab plus nivolumab

INTERVENTIONS:
Drug: Ipilimumab plus nivolumab plus guadecitabine — Cohort A Melanoma ARM A Guadecitabine: 30-45 mg/m2 s.c./day 1-5 q21 x 4 cycles and from W13 q28 x 6 cycles Ipilimumab: 3 mg/Kg i.v. plus nivolumab 1 mg/Kg i.v. on W1, 4, 7 and 10 and from W14 nivolumab 480 mg i.v. q4 wks for 2 years
  Cohort B NSCLC ARM A Guadecitabine: 30-45 mg/m2 s.c./day 1-5 q21 x 4 cycles and from W13 q28 x 6 cycles Ipilimumab: 1 mg/Kg i.v.q 6wks plus nivolumab 3 mg/Kg i.v. q2 wks until W13, then ipilimumab: 1 mg/Kg i.v. q 6wks plus nivolumab 480mg i.v. q4wks for 2 years
  Other Names: ipilimumab (Yervoy); nivolumab (Opdivo); guadecitabine (SGI-110)
  Arms: Ipilimuamb plus nivoluamb plus guadecitabine
Drug: Ipilimumab plus nivolumab — Cohort A Melanoma ARM B Ipilimumab: 3 mg/Kg i.v. plus nivolumab 1 mg/Kg i.v. on W1, 4, 7 and 10 and from W14 nivolumab 480 mg i.v. q4 wks for 2 years
  Cohort B NSCLC ARM B Ipilimumab: 1 mg/Kg i.v. q 6wks plus nivolumab 3 mg/Kg i.v. q2 wks until W13, then ipilimumab: 1 mg/Kg i.v. q6 wks plus nivolumab 480mg i.v. q4wks for 2 years.
  Other Names: ipilimumab (Yervoy); nivolumab (Opdivo)
  Arms: Ipilimumab plus nivolumab

SUMMARY:
This is a run-in, randomized, non-comparative, phase II study designed according to a two stages optimal design by Simon. This phase II design will be preceded by a safety evaluation after the first cohort of 6 patients to preserve a high-grade of overlapping and/or unexpected toxicity rate. The study will assess the immune-objective response rate (iORR) (assessed using iRECIST criteria) of nivolumab combined with ipilimumab and guadecitabine or nivolumab combined with ipilimumab, in Melanoma and non-small cell lung cancer (NSCLC) patients resistant to anti-PD-1/PD-L1 therapy. Immune biologic correlates to treatment will be assessed as exploratory endpoints.

DETAILED DESCRIPTION:
Epigenetic alterations play a pivotal role in cancer development and progression. Pharmacologic reversion of such alterations is feasible, second generation "epigenetic drugs" are in development and have demonstrated to possess significant immunomodulatory properties. This knowledge, together with the availability of new and highly effective immuno-therapeutic agents including immune check-point(s) blocking monoclonal antibodies, allows the investigators to plan for highly innovative proof-of-principle combination studies that will likely open the path to more effective anti-cancer therapies. Targeting immune check-point(s) with immunomodulatory monoclonal-antibodies is a novel and rapidly evolving strategy to treat cancer, that is rapidly spreading to different tumor histologies. The prototype approach of this therapeutic modality relies on the inhibition of negative signals delivered by CTLA-4 expressed on T lymphocytes. CTLA-4 blockade has profoundly changed the therapeutic landscape of melanoma, significantly improving the survival of patients; however, objective clinical responses are limited, and only a minority of patients achieves long-term disease control. Therefore, several combination approaches are being explored to improve the efficacy of CTLA-4 blockade. The anti-PD-1 monoclonal antibodies, nivolumab and pembrolizumab, have significantly increased the survival of melanoma and NSCLC patients. Despite this unprecedented efficacy, a significant proportion of melanoma and NSCLC patients fails to respond (primary resistance) or develops secondary resistance to anti-PD-1 treatment over time. Therefore, identifying new mechanism(s) underlying treatment failure(s), and designing novel combination/sequencing therapeutic approaches to overcome primary/secondary resistance is mandatory to improve the overall efficacy of anti-PD-1 therapy. The investigators have first demonstrated that epigenetic immune-modeling of cancer cells represents a key hallmark of cancer, as it impairs functional host's immune recognition of malignant cells; on the other hand, the investigators have shown the potential of epigenetic drugs, including DNA hypomethylating agents (DHA), to sensitize tumor cells to emerging immunotherapies. Based on these pre-clinical in vitro and in vivo findings, the investigators have most recently promoted the clinical translation of the immunomodulatory potential of epigenetic drugs through highly-innovative, hypothesis-driven, clinical trials. Along this line, the ongoing, exploratory, Investigator Initiated Trial (IIT) phase Ib NIBIT-M4 study, has evaluated safety and immunobiologic activities of the epigenetic priming with the next generation DHA guadecitabine followed by CTLA-4 blockade in MM patients (NCT02608437). The results of NIBIT-M4 study support the notion that DHA represent ideal "partner drugs" to improve the therapeutic efficacy of immune-checkpoint blockade, including the foreseeable role in reverting resistance to treatment. The NIBIT-ML1 study will assess the therapeutic efficacy of nivolumab combined with ipilimumab and guadecitabine or nivolumab combined with ipilimumab, in metastatic melanoma and NSCLC patient with primary resistance to anti-PD-1/PD-L1 therapy. Exploratory translational objectives will extensively investigate, on neoplastic cells, tumor microenveroinment and peripheral blood, immune-biologic correlates to treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Target Population Melanoma cohort A

   1. Histologic diagnosis of malignant melanoma
   2. Unresectable Stage III/Stage IV melanoma patients with resistance to anti-PD-1/PD-L1 and measurable lesions by CT or MRI per iRECIST/RECIST criteria that can be amenable to biopsy
   3. Only one line of immunotherapy for advanced (unresectable Stage III or Stage IV) disease with anti-PD-1/PD-L1 and its combinations; if BRAF mutant one line of targeted therapy is allowed prior to anti-PD-1/PD-L1therapy.
2. Target Population NSCLC cohort B

   1. Histologic or cytologic diagnosis of NSCLC lackingEGFR-sensitizing mutation and/or ALK/ROS1 translocation.
   2. Stage IV NSCLC patients with primary resistance to anti-PD-1/PD-L1 and measurable lesions by CT or MRI per iRECIST/RECIST criteria that can be amenable to biopsy.
   3. Only one line of immunotherapy for advanced (unresectable Stage III or Stage IV) disease with anti-PD-1/PD-L1 or its combinations; one line of chemotherapy is allowed prior to anti-PD-1/PDL-1 therapy.
3. confirmed PD
4. 4 weeks or greater since last treatment and
5. Must have recovered from any acute toxicity associated with prior therapy
6. Life expectancy greater than 16 weeks
7. Subjects with adequate organ function defined as:

   1. WBC ≥3500/uL
   2. ANC ≥2000/uL
   3. Platelets ≥ 100 x 103/uL
   4. Hemoglobin ≥ 9 g/dL
   5. Creatinine < or <= 2.5 x ULN
   6. AST

      * < or <= 2.5 x ULN for patients without liver metastasis
      * < or <= 5 x ULN for patients with liver metastasis
   7. Bilirubin

      * < or <= 3 x ULN for patients with liver metastasis
      * <3.0 mg/mL for patients with Gilbert's Syndrome
      * 1.5 x ULN for patients without liver metastasis
8. Negative screening tests for HIV, HepB, and HepC. If positive results are not indicative of true active or chronic infection, the patient can enter the study after discussion and agreement between the Investigator and the Medical Monitor.
9. Women of child-bearing potential must not be pregnant or breastfeeding, must have a negative pregnancy test at Screening and all men must be practicing two medically acceptable methods of birth control. Men should not father a child while receiving treatment with guadecitabine+ ipilimumab, and for 2 months following completion of treatment. Men with female partners of childbearing potential should use effective contraception during this time.

Exclusion Criteria:

1. Sex and Reproductive Status

   1. Women who are pregnant or breastfeeding;
   2. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 23 weeks after the study;
   3. Women with a positive pregnancy test on enrollment or prior to investigational product administration;
   4. Sexually active fertile men not using effective birth control if their partners are WOCBP
2. Target Disease Exceptions

   1. Any malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix
   2. Primary ocular melanoma.
3. Medical History and Concurrent Diseases

   1. Symptomatic brain metastases requiring immediate local intervention (radiotherapy (RT) and/or surgery);
   2. Leptominingeal involvement by disease;
   3. Autoimmune disease: Patients with a documented history of Inflammatory Bowel Disease, including ulcerative colitis and Crohn's disease are excluded from this study as are patients with a documented history of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis] and autoimmune hepatitis. Subjects with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre Syndrome) are also excluded from this study;
   4. Any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
4. Prohibited Treatments and/or Therapies

   1. Concomitant therapy with any anti-cancer agent; immunosuppressive agents; any non-oncology vaccine therapy used for prevention of infectious diseases (for up to 1 month prior to or after any dose of study drug); surgery or radiotherapy (except palliative surgery and/or radiotherapy to treat a non-target symptomatic lesion or to the brain after Sponsor approval); other investigational anti-cancer therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses);
   2. Previous treatment with other investigational products, including cancer immunotherapy, within 30 days;
   3. Prior treatment with anti-CTLA-4, except in adjuvant setting Other Exclusion Criteria

   <!-- -->

   1. Prisoners or subjects who are involuntarily incarcerated;
   2. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Eligibility criteria for this study have been carefully considered to ensure the safety of the study subjects and to ensure that the results of the study can be used. It is imperative that subjects fully meet all eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Immune-related Objective Response Rate (iORR) | 24 weeks
  Immune-related Objective Response Rate (iORR) is the proportion of treated subjects with an iBOR of confirmed iCR or confirmed iPR.

SECONDARY OUTCOMES:
Safety of guadecitabine in combination with ipilimumab and nivolumab | 2 years
  Reporting of safety, extent of exposure, concomitant medications and discontinuation of study therapy will be based on all treated subjects; for on-study laboratory test results, all treated subjects with at least one on-study laboratory measurement available will be included in the analysis. The reporting period for safety data will be from the date of first dose received on this study to 100 days after the last dose is received. Serious adverse events are reported from the time of consent forward for all subjects. All subjects who received at least one dose of study treatment will be evaluated for safety parameters
Obiective Response Rate (ORR) | 24 weeks
  Objective Response Rate (ORR) is the proportion of treated subjects with a BOR of CR or PR per RECIST 1.1.
Disease Control Rate (DCR) | 24 weeks
  Disease Control Rate (DCR) is the proportion of treated subjects with a BOR of confirmed CR, confirmed PR or SD, based on RECIST 1.1 and iRECIST.
Duration of response (DoR) | 2 years
  Duration of Response (DoR) for the subjects whose BOR is CR or PR will be defined as the time between the date of response of confirmed CR or confirmed PR (whichever occurs first) and the date of PD or death (whichever occurs first), based on RECIST 1.1 and iRECIST.
Time to response (TTR) | 24 weeks
  Time to Response (TTR) is defined as the time from first dosing date until the measurement criteria are first met for overall response of PR or CR (whichever status comes first, and provided it is subsequently confirmed), , based on RECIST 1.1 and iRECIST.
Progression Free Survival (PFS) | 2 years
  Progression free survival (PFS) per RECIST 1.1 and iRECISTwill be defined as the time between the date of randomization and the date of progression and or confirmed PD (according to RECIST 1.1 and iRECIST) or death, whichever occurs first.
Overall Survival (OS) | 2 years
  Overall Survival (OS) is defined as the time from randomization until the date of death. For those subjects who have not died, OS will be censored at the recorded last date of subject contact, and for subjects with a missing recorded last date of contact, OS will be censored at the last date the subject was known to be alive. Any efforts will be made to know the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Di Giacomo, MD, Principal Investigator — Center for Immuno-Oncology, University Hospital of Siena
Locations (1):
- Center for Immuno-Oncology, University Hospital of Siena, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Larkin J, Hodi FS, Wolchok JD. Combined Nivolumab and Ipilimumab or Monotherapy in Untreated Melanoma. N Engl J Med. 2015 Sep 24;373(13):1270-1. doi: 10.1056/NEJMc1509660. No abstract available. PMID 26398076
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Maio M, Di Giacomo AM, Robert C, Eggermont AM. Update on the role of ipilimumab in melanoma and first data on new combination therapies. Curr Opin Oncol. 2013 Mar;25(2):166-72. doi: 10.1097/CCO.0b013e32835dae4f. PMID 23299197
- [Background] Maio M, Covre A, Fratta E, Di Giacomo AM, Taverna P, Natali PG, Coral S, Sigalotti L. Molecular Pathways: At the Crossroads of Cancer Epigenetics and Immunotherapy. Clin Cancer Res. 2015 Sep 15;21(18):4040-7. doi: 10.1158/1078-0432.CCR-14-2914. PMID 26374074
- [Background] Sigalotti L, Fratta E, Coral S, Maio M. Epigenetic drugs as immunomodulators for combination therapies in solid tumors. Pharmacol Ther. 2014 Jun;142(3):339-50. doi: 10.1016/j.pharmthera.2013.12.015. Epub 2013 Dec 30. PMID 24384533
- [Background] Di Giacomo AM, Covre A, Finotello F, Rieder D, Danielli R, Sigalotti L, Giannarelli D, Petitprez F, Lacroix L, Valente M, Cutaia O, Fazio C, Amato G, Lazzeri A, Monterisi S, Miracco C, Coral S, Anichini A, Bock C, Nemc A, Oganesian A, Lowder J, Azab M, Fridman WH, Sautes-Fridman C, Trajanoski Z, Maio M. Guadecitabine Plus Ipilimumab in Unresectable Melanoma: The NIBIT-M4 Clinical Trial. Clin Cancer Res. 2019 Dec 15;25(24):7351-7362. doi: 10.1158/1078-0432.CCR-19-1335. Epub 2019 Sep 17. PMID 31530631
- [Background] Covre A, Coral S, Di Giacomo AM, Taverna P, Azab M, Maio M. Epigenetics meets immune checkpoints. Semin Oncol. 2015 Jun;42(3):506-13. doi: 10.1053/j.seminoncol.2015.02.003. Epub 2015 Feb 14. PMID 25965370
- [Background] Hodi FS, Chiarion-Sileni V, Gonzalez R, Grob JJ, Rutkowski P, Cowey CL, Lao CD, Schadendorf D, Wagstaff J, Dummer R, Ferrucci PF, Smylie M, Hill A, Hogg D, Marquez-Rodas I, Jiang J, Rizzo J, Larkin J, Wolchok JD. Nivolumab plus ipilimumab or nivolumab alone versus ipilimumab alone in advanced melanoma (CheckMate 067): 4-year outcomes of a multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Nov;19(11):1480-1492. doi: 10.1016/S1470-2045(18)30700-9. Epub 2018 Oct 22. PMID 30361170
- [Background] Ready N, Hellmann MD, Awad MM, Otterson GA, Gutierrez M, Gainor JF, Borghaei H, Jolivet J, Horn L, Mates M, Brahmer J, Rabinowitz I, Reddy PS, Chesney J, Orcutt J, Spigel DR, Reck M, O'Byrne KJ, Paz-Ares L, Hu W, Zerba K, Li X, Lestini B, Geese WJ, Szustakowski JD, Green G, Chang H, Ramalingam SS. First-Line Nivolumab Plus Ipilimumab in Advanced Non-Small-Cell Lung Cancer (CheckMate 568): Outcomes by Programmed Death Ligand 1 and Tumor Mutational Burden as Biomarkers. J Clin Oncol. 2019 Apr 20;37(12):992-1000. doi: 10.1200/JCO.18.01042. Epub 2019 Feb 20. PMID 30785829
- [Background] Lebbe C, Meyer N, Mortier L, Marquez-Rodas I, Robert C, Rutkowski P, Menzies AM, Eigentler T, Ascierto PA, Smylie M, Schadendorf D, Ajaz M, Svane IM, Gonzalez R, Rollin L, Lord-Bessen J, Saci A, Grigoryeva E, Pigozzo J. Evaluation of Two Dosing Regimens for Nivolumab in Combination With Ipilimumab in Patients With Advanced Melanoma: Results From the Phase IIIb/IV CheckMate 511 Trial. J Clin Oncol. 2019 Apr 10;37(11):867-875. doi: 10.1200/JCO.18.01998. Epub 2019 Feb 27. PMID 30811280
- See also: Fondazione NIBIT Onlus Network Italiano per la Bioterapia dei Tumori — http://fondazionenibit.org